CLINICAL TRIAL: NCT04146337
Title: Fecal Microbiota Transplantation for Eradication of Carbapenem-resistant Enterobacteriaceae Colonization: Randomized Control Trial
Brief Title: Fecal Microbiota Transplantation for Carbapenem-resistant Enterobacteriaceae
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0338-19
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Carbapenem-Resistant Enterobacteriaceae Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal microbiota transplantation (FMT) (Experimental): FMT regimen: Patients will be given capsulized FMT 15 capsules a day for two consecutive days after a fast of 8 hours before FMT. Stool will be collected before and after the intervention for genomic analysis of CRE strains, analysis of microbiome and metabolome.
  Interventions: Biological: FMT
- Control (No Intervention): Routine follow-up

INTERVENTIONS:
Biological: FMT — Fecal microbiota in frozen capsules
  Arms: Fecal microbiota transplantation (FMT)

SUMMARY:
2:1, open-label, single center, randomized controlled trial comparing FMT vs. no intervention for CRE carriers,

DETAILED DESCRIPTION:
Antibiotic resistance has emerged worldwide and is of major concern leading to multidrug resistant (MDR) bacteria that are widely spread and are a major factor in morbidity and mortality in health-care settings. Among MDRs, carbapenem resistant Enterobacteriaceae (CRE) are of special concern, receiving the highest classification of "urgent threat level" in the US President Report. Consistent mortality rates of 40-50% are observed among inpatients with infections caused by CRE in hospitals worldwide, related mainly to unavailable, delayed or ineffective antibiotic treatment options. The extremely high mortality rates of patients with CRE infections have driven efforts to prevent the acquisition and spread of these bacteria in hospitals. These include screening for carriage, contact isolation of carriers, cohorting, dedicated healthcare staff and other infection control measures. These strategies have been proven as effective but are cumbersome and expensive. In most locations these strategies failed to completely eradicate CRE endemicity. CRE decolonization (eradication of colonization) might offer a double benefit: reducing the risk for the individual carrier to develop an infection due to the resistant strain (by that, potentially lowering the mortality risk) and preventing the bacteria from spreading to other patients, exposing them to the same hazard. Fecal microbiota transplantation (FMT), in which fecal material enriched with commensal microorganisms is transferred from a healthy donor, have proven efficacy in the treatment of recurrent Clostridium difficile infection (CDI) in multiple trails. Major adverse events that has been reported so far are mostly related to the route of administration (aspiration during nasogastric tube administration/colonoscopy). Other adverse events include mostly GI related symptoms (diarrhea, nausea, belching) and are self limited and resolve in few hours. FMT seems to be safe and effective both in immunocompetent and immunocompromised patients. The high efficacy of FMT in the treatment of a multi-drug resistant pathogen such as Clostridium difficile, suggest that it might be an efficient tool for other MDR pathogens (e.g. CRE). The potential of FMT to restore the gut microbiome and compete with residual resistant strains offer a novel way to fight the current MDR epidemic.

The investigators aim to assess the effects of FMT on colonization and clinical infections with CRE. The investigators will apply FMT on a cohort of CRE carriers in a single center in Israel. FMT will be given by capsules for 2 consecutive days followed by rectal sampling at predefined time-point in the following 6 months.

ELIGIBILITY:
We will include adult inpatients ≥18 years positive for CRE of any strain and resistance mechanism in rectal surveillance stool samples, with or without CRE clinical samples. We will mandate a positive rectal swab within one week before randomization. Several exclusion criteria may change throughout the patients' hospitalization and we will follow-up patients for these criteria until reaching eligibility or not (designed as (for follow-up)). Non-eligible patients discharged will be re-evaluated for inclusion when re-admitted.

We will exclude:

* Pregnant women
* Patients with severe neutropenia (<100/µl) (for follow-up)
* Severe GVHD involving the gastrointestinal involvment (for follow-up)
* Patients with inflammatory bowel disease (Crohn's or ulcerative colitis)
* Patients with intestinal perforation or severe abdominal infection (for follow-up)
* Patients carrying a colostomy, ileostomy or similar
* Inability or contra-indication to take oral medications (intestinal obstruction, suspected perforation, peritonitis) (for follow-up)
* Severe food allergies
* Severe diarrhea (for follow-up)
* Inability to provide informed consent (for follow-up)
* Refusal of primary care physician
* Patients treated with antibiotics within the 2 days before fulfilling all other eligibility criteria (for follow-up)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
CRE eradication | 28 days
  Number of participants achieving CRE eradication at 28 days, defined as 3 consecutive negative rectal cultures, with polymerase chain reaction preformed in the last sample. For patients with clinical infections, eradication definition will include a negative culture from the site of infection, if relevant at the time of eradication.

SECONDARY OUTCOMES:
CRE eradication rates at day 7, day 14, and 3 & 6 months | days 7, 14, months 3, 6
  Number of participants achieving CRE eradication rates at day 7, day 14, and 3 & 6 months
Mortality | 28-day and 6 months
  Number of participants who died by 28-day and 6 month
Bacteremia | 6 months
  Number of participants with CRE bacteremia and any bacteremia
CRE infection | 6 months
  Number of participants with non-bacteremic new clinically-significant CRE infections
Hospitalization days | 6 months
  Totals days in-hospital
Adverse events | 6 months
  Number of participants with: pneumonia within a week after the intervention; dyspeptic complaints collected at the time of rectal sampling; changes in bowel habit including diarrhea and constipation; discontinuation of FMT before completing the study protocol

CONTACTS AND LOCATIONS:
Overall Officials: Haggay Bar Yoseph, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Yes
Share by contact with authors
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: End of study
Access Criteria: Academic use